CLINICAL TRIAL: NCT06257797
Title: Fenugreek: New Therapeutic Resource or Emerging Allergen
Brief Title: Fenugreek: an Emergent Allergen
Status: Completed | Type: Observational
Sponsor: Paola Miciullo (Other)
Responsible Party: Sponsor-Investigator, Paola Miciullo, Associated Professor, Azienda Ospedaliera Universitaria Policlinico "G. Martino"
Organization: Azienda Ospedaliera Universitaria Policlinico "G. Martino" (Other)
Other Study IDs: 3/24
Record Dates: First submitted 2024-02-01; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Fenugreek Hypersensitivity - Cross-reactivity - Food Allergy
MeSH Terms: interventions — Patch Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Allergic patients to fenugreek
  Interventions: Diagnostic Test: Skin prick test
- Non allergic patients to fenugreek
  Interventions: Diagnostic Test: Skin prick test

INTERVENTIONS:
Diagnostic Test: Skin prick test — Fenugreek wiil be tested by mixing fenugreek seed powder with saline at non-irritating doses and it will be performed by prick-by-prick test. The skin tests will be read 20 minutes after the execution.

SUMMARY:
Fenugreek or Trigonella foenum greacum is an ancient medicinal plant native to the eastern Mediterranean, later spread to Asia (especially in India); it belongs to Rosaceae order, Leguminosae family, subfamily of Papilonaceae and it is used as a medicinal herb, spice or food. It is a component of spice mix, such as curry, and it is also used as a supplement in wheat and corn flour for bread-making. Fenugreek appears to have many health benefits and potential medicinal properties (antioxidant, antidiabetic, hepatoprotective, hypocholesterolemic, antimicrobial, anti-inflammatory, neuroprotective, anticarcinogenic, antiulcer, and antilithigenic) both in vitro and in vivo studies; for this reason it may be increasingly being used as nutraceutical formulations (powder, herbal teas, tablets and various combinations).This study aims to describe patients who came to our operating unit for suspected adverse reaction after ingestion of fenugreek and to highlight possible cross-reactivity between fenugreek and other legumes or other foods. Given the increasing use of novel spices in Mediterranean cuisine and the possible spread of fenugreek-based nutraceuticals, it is relevant to draw attention to possible allergic reactions.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 yo
* history of allergic reactions to spices
* history of allergic reactions to phytotherapics containing fenugreek

Exclusion Criteria:

* age < 18 yo
* non suggestive history of allergic reactions to spices

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients referred to outpatients visit to the Operative Unit of Allergy and Clinical Immunology of Messina University Hospital with a suggestive history of allergy after ingestion of spices and tested for fenugreek.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Cutaneous sensitization to fenugreek | 1 hour
  Cutaneous sensitization to fenugreek evaluated by the result of skin prick test in patients with suggestive history of allergic reactions to spices.

SECONDARY OUTCOMES:
Cross-reactivity between fenugreek and other legumes and other foods | 1 hour
  Cutaneous sensitization to other legumes (lentil, bean, pea, soy, lupine and peanut) and other foods evaluated by the result of skin prick test in patients with suggestive history of allergic reactions to spices.

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Policlinico Universitario G. Martino, Messina, Sicily/Messina, Italy

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-15): https://cdn.clinicaltrials.gov/large-docs/97/NCT06257797/Prot_SAP_000.pdf
  • Informed Consent Form (2024-01-15): https://cdn.clinicaltrials.gov/large-docs/97/NCT06257797/ICF_001.pdf